# Technical Trial Statistical Analysis Plan-CTR display plan

# **AERIAL®**

Changes in health and functional status in patients with COPD during therapy with Spiolto<sup>®</sup> Respimat<sup>®</sup>

Project No: 5312000\_AERIAL

Medication: Spiolto® Respimat®

**Dokument ID:** TechnicalSAP\_1237-0065\_Final\_3.0\_2019-03-12.docx

**Version:** Final 3.0 **Date:** 12.03.2019

Sponsor: Boehringer Ingelheim International GmbH

Binger Straße 173

55216 Ingelheim am Rhein

Germany

**Author:** 

Protocol (Version, Date): Version 2.0, 24.04.2017

#### Tables of contents

| 1 M | ethods for calculat | ion of derived variables | 3 |
|---|---|---|---|
| 2 D | ISPLAY TEMPLAT | ES | 5 |
| 2.1 | Display templat | es for in - text reports | 5 |
| 2. | 1.1 In-text table ter | mplates | 5 |
| 2. | 1.1 In-text figur | re examples | 5 |
| 2.2 | Display templat | es for in- or end-of-text reports | 5 |
| 2. | 2.1 End-of-text | table templates | 5 |
| | 2.2.1.1 15.1 | Trial subject | 5 |
| | 2.2.1.1.1 15 | 5.1.1 Disposition of subjects | 5 |
| | 2.2.1.1.2 15 | 5.1.3 Definition of analysis sets | 7 |
| | 2.2.1.1.3 15 | 5.1.4 Demographic data and baseline characteristics | 7 |
| | 2.2.1.1.4 15 | 5.2. Efficacy evaluation | 20 |
| | 2.2.1.1.5 15 | 5.3. Safety analysis | 23 |
| 2.3 | Sensitivity analy | ysis I- Time between Visit 1 and Visit 2 | 30 |
| 2.4 | Sensitivity analy | ysis II- Non-estimated number of exacerbations* | 32 |
| 2.5 | Tables for subg | roup analysis | 36 |
| 2.6 | Appendix | | 41 |
| 2.7 | Listings | | 44 |

The following tables, listings and figures are planned. The checkered fields as well as the terms in brackets {...} show the programmer where the parameter to be analysed may be found and will not appear in the report. In this context, the variable before the point displays the dataset and the variable after the point stands for the field name within the corresponding dataset. Take note, that the variable before the point must be always reported again as first term after the point, e.g. patient.birthyear stands for the field patient.patient\_birthyear in the eCRF.

#### 1 Methods for calculation of derived variables

<u>Age at registration:</u> Year of registration {year(registration.registered\_at)} - Year of birth {patient.birthyear}

Clinical COPD Questionnaire (CCQ): Each of the 10 CCQ questions is scored by the patient on a 7-point scale between 0 (Never/Not limited at all) and 6 (Almost all the time/Totally limited or unable to do) at baseline and end of the observation after approximately 6 weeks. The (total) CCQ score measures the health and functional status. A higher CCQ score is indicative of worse status and a decrease of 0.4 points is considered to be the minimum clinically important difference (MCID). The total CCQ score and the corresponding subscales are calculated as followed, in case that at least the number of required answers is available:

| Scale | Items | Items required | Scoring<br>(For details see www.ccq.nl) | Field names |
|---|---|---|---|---|
| Symptom | 1; 2; 5;<br>6 | 3 | Sum of answered questions Number of answered questions | ccq.q_<br>[01;02;05;06] |
| Functional state (CCQ-4) | 7-10 | | Sum of answered questions Number of answered questions | ccq.q_07-<br>ccq.q_10 |
| Mental state 3; 4 2 | | 2 | $\frac{Item\ 3+4}{2}$ | ccq.q_03;<br>ccq.q_04 |
| Total CCQ score | | ales must<br>culable | $\frac{(Symptom + Functional state)*4 + (Mental state)*2}{10}$ | ccq.q_01-<br>ccq.q_10 |

<u>Change of CCQ score:</u> total CCQ score at baseline minus total CCQ score after approximately 6 weeks

<u>Therapeutic success:</u> total CCQ score at baseline minus total CCQ score after approximately 6 weeks is greater or equal to 0.4

Non therapeutic success: total CCQ score at baseline minus total CCQ score after approximately 6 weeks is less than 0.4

<u>Share of patients with therapeutic success:</u> number of patients with therapeutic success divided by total number of patients

#### mMRC questionnaire {mmrc.activity}:

| mMRC Classification | Answer |
|---|---|
| Grade 0 | Breathless with strenuous exercise |
| Grade 1 | Short of breath when hurrying on the level or walking up a slight hill |
| Grade 2 | Walk slower than people of the same age on the level because of breathlessness, or have to stop for breath when walking at own pace on the level |
| Grade 3 | Stop for breath after walking about 100 meters or after a few minutes on level |
| Grade 4 | Too breathless to leave the house or breathless when dressing or undressing |

Final 3.0, 12.03.2019 3 / 53

#### **GOLD** group

| GOLD<br>group | Definition | Exacerbations* per year {anamnesis.exacerbation} and/or hospitalizations due to excerbations {anamnesis_exacerbation_hospital} | mMRC<br>classification<br>{mmrc.activity} |
|---|---|---|---|
| Α | | 0-1 and =0 | ≤1 |
| В | Low risk, more symptoms | 0-1 and =0 | ≥ 2 |
| С | High risk , less symptoms | ≥ 2 or ≥1 | 0-1 |
| D | High risk , more symptoms | ≥ 2 or ≥1 | ≥ 2 |

<sup>\*</sup>For unknown number of exacerbations "0" is included in the calculation of the GOLD group

If 0 or 1 excerbation per year is documented along with a mMRC of at least grade 2 at baseline the patient is assigned GOLD group B.

If two and more excerbations per year are documented along with a mMRC of grade 0 or 1 at baseline the patient is assigned GOLD group C.

If two and more excerbations per year are documented along with a mMRC of at least grade 2 at baseline the patient is assigned GOLD group D.

<u>Duration between initial diagnosis of COPD and baseline visit:</u> Year of Visit 1 {year(anamnesis.date)}- Year of initial COPD diagnosis {anamnesis.copd\_year}

<u>Time between start of treatment and end of observation/discontinuation [weeks]:</u> (Date of Visit 2 {visit.date}/Date of last treatment within observation period {visit.spiolto\_last\_date}-Date of start of treatment {anamnesis.spiolto\_date})/7

<u>Time between Visit 1 and Visit 2 [weeks]:</u> (Date of Visit 2 {visit.date}-Date of Visit 1 {anamnesis.date})/7

<u>Pack years:</u> (Years of smoking)\*(Cigarette parcels per day){anamnesis.smoker\_pack\_years; visit.smoker\_pack\_years}

Final 3.0, 12.03.2019 4 / 53

#### **2 DISPLAY TEMPLATES**

### 2.1 Display templates for in - text reports

## 2.1.1 In-text table templates

Not applicable.

### 2.1.1 In-text figure examples

Not applicable.

### 2.2 Display templates for in- or end-of-text reports

### 2.2.1 End-of-text table templates

#### 2.2.1.1 15.1 Trial subject

# **2.2.1.1.1 15.1.1 Disposition of subjects**

Table 15.1.1 1: Disposition

| | N (%) |
|---|---|
| Patients recruited {patient.id} | xx (100.0) |
| Patients with visit 1 {anamnesis.done} | xx (yy.y) |
| Reason for not performing Visit 1 {anamnesis.done_reason} | (333) |
| Adverse event | xx (yy.y) |
| Serious adverse event | xx (yy.y) |
| Patient's wish | xx (yy.y) |
| Withdrawn consent | xx (yy.y) |
| Lost to follow-up | xx (yy.y) |
| Patient died | xx (yy.y) |
| Other | xx (yy.y) |
| Study participation not possible {patient.no_participation} | xx (yy.y) |
| Patients with visit 1, but no registration {anamnesis.done}{registration.registered_by} | xx (yy.y) |
| Patients not treated | xx (yy.y) |
| Patients included in Treated Set | xx (yy.y) |
| Patients with Visit 2 {visit.done} | |
| Reason for not performing Visit 2 {visit.done_reason} | xx (yy.y) |
| Adverse event | xx (yy.y) |
| Serious adverse event | xx (yy.y) |
| Patient's wish | xx (yy.y) |
| Withdrawn consent | xx (yy.y) |
| Lost to follow-up | xx (yy.y) |
| Patient died | xx (yy.y) |
| Other | xx (yy.y) |
| Patients with Visit 2- Continuation of medication after end of observation (Spiolto <sup>®</sup> Respimat <sup>®</sup> ) {visit.spiolto_continued} | xx (yy.y) |
| Patients with Visit 2- Discontinuation of medication after end of observation (Spiolto <sup>®</sup> Respimat <sup>®</sup> ) | xx (yy.y) |
| Reason for discontinuation of Spiolto® Respimat® {visit.spiolto_reason} | |
| Adverse event | xx (yy.y) |
| Serious adverse event | xx (yy.y) |
| Patient's wish | xx (yy.y) |
| Withdrawn consent | xx (yy.y) |
| Lost to follow-up | xx (yy.y) |
| Patient died | xx (yy.y) |
| Other | xx (yy.y) |

Final 3.0, 12.03.2019 5 / 53

| Patients included in FAS | xx (yy.y) |
|-------------------------------------------|-----------|
| Reason for not included in FAS | |
| Available total CCQ score at visit 1 only | xx (yy.y) |
| Available total CCQ score at visit 2 only | xx (yy.y) |
| No available total CCQ score at all | xx (yy.y) |
| Not included in TS | xx (yy.y) |

#### 15.1.2 Important protocol violations

### Table 15.1.2 1: Patients with visit 1- Important protocol violations

| | N (%) |
|---|---|
| Total | xx (100.0) |
| Total with violation of informed consent {patient.ic_01} | xx (yy.y) |
| Total with violation of any other inclusion criteria {patient.ic_02-patient.ic_04} | xx (yy.y) |
| Total with violation of any exclusion criteria {patient.ec_01-patient.ec_05} | xx (yy.y) |
| Total with violation of any inclusion or exclusion criteria { patient.ic_01-patient.ic_04; patient.ec_01-patient.ec_05} | xx (yy.y) |

#### Table 15.1.2 2 Patients with visit 1- Inclusion criteria

| Inclusion criteria not fulfilled | N | % |
|---|---|---|
| patient.ic_01 | | |
| IC 1- Written informed consent prior to participation | | |
| patient.ic_03 | | |
| IC 2- Female and male patients >=40 years of age | | |
| patient.ic_02 | | |
| IC 3- Patients diagnosed with COPD and requiring a combination of two longacting bronchodilators (LAMA+LABA) according to approved SmPC and GOLD COPD guideline recommendation 2017 (GOLD COPD groups B to D) | | |
| patient.ic_04 | | |
| IC 4- Treatment with Spiolto <sup>®</sup> Respimat <sup>®</sup> acc. to SmPC at the discretion of the physician | | |
| At least one inclusion criteria not fulfilled | | |
| Number of patients | XX | 100.00 |

### Table 15.1.2 3: Patients with visit 1- Exclusion criteria

| Exclusion criteria fulfilled | N | % |
|---|---|---|
| patient.ec_01 | | |
| EC 1- Patients with contraindications according to Spiolto® Respimat® SmPC | | |
| patient.ec_02 | | |
| EC 2- Patients already on a LABA/LAMA combination (free and fixed dose) in the last 6 weeks before study entry | | |
| patient.ec_03 | | |
| EC 3- Patients continuing LABA-ICS treatment should not be additionally treated with Spiolto <sup>®</sup> Respimat <sup>®</sup> in order to avoid a double dosing of long-acting beta-agonists | | |

Final 3.0, 12.03.2019 6 / 53

| Exclusion criteria fulfilled | N | % |
|---|---|---|
| patient.ec_05 | | |
| EC 4- Pregnancy and lactation | | |
| patient.ec_04 | | |
| EC 5- Current participation in any clinical trial or any other non-interventional study of a drug or devise | | |
| At least one exclusion criteria fulfilled | | |
| Number of patients | xx | 100.00 |

### 2.2.1.1.2 15.1.3 Definition of analysis sets

Table 15.1.3 1: Patients with visit 1 patients- Summary of analysis population

| Sample size | N | % |
|-------------------------|----|--------|
| Treated Set (TS) | | |
| Full Analysis Set (FAS) | | |
| Patients with visit 1 | XX | 100.00 |

### 2.2.1.1.3 15.1.4 Demographic data and baseline characteristics

Table 15.1.4 1: Treated Set- Age at registration [years]

| patient.birthyear;<br>registration.registered_at | N<br>(Number of non-<br>missing values) | Mean | SD | Min | Median | Max | Nmiss<br>(Number of<br>missing values) |
|---|---|---|---|---|---|---|---|
| Age at registration | | | | | | | |

Table 15.1.4 2: Treated Set- Age at registration, categorical

| | 9.00. | , |
|--------------------------------------------------|-------|---|
| patient.birthyear;<br>registration.registered_at | N | % |
| Age, categorical | | |
| <65 years | | |
| ≥65 years | | |
| Missing | | |
| Number of patients | | |

Table 15.1.4 3: Treated Set- Gender

| patient.gender<br>Gender | N | % |
|--------------------------|---|---|
| Male | | |
| Female | | |
| Number of patients | | |

Final 3.0, 12.03.2019 7 / 53

#### Table 15.1.4 4: Treated Set- Height [cm]

| patient.bodysize | N | Mean | SD | Min | Median | Max | Nmiss |
|------------------|---|------|----|-----|--------|-----|-------|
| Height | | | | | | | |

#### Table 15.1.4 5: Treated Set- Weight [kg]

| patient.bodyweight | Ν | Mean | SD | Min | Median | Max | Nmiss |
|--------------------|---|------|----|-----|--------|-----|-------|
| Weight | | | | | | | |

#### Visit 1- Baseline

# Table 15.1.4 6: Treated Set- Duration between initial diagnosis of COPD and baseline visit [years]

| anamnesis.date; anamnesis.copd_year | N | Mean | SD | Min | Median | Max | Nmiss |
|---|---|---|---|---|---|---|---|
| Duration between initial diagnosis and baseline visit | | | | | | | |

#### Table 15.1.4 7: Treated Set- COPD degree of severity (spirometric)

| anamnesis.copd_severity | N | % |
|---------------------------------------|----|----|
| COPD degree of severity (spirometric) | 11 | 70 |
| 1 | | |
| 2 | | |
| 3 | | |
| 4 | | |
| No preliminary examination result | | |
| Missing | | |
| Number of patients in Treated Set | | |

#### Table 15.1.4 8: Treated Set- COPD degree of severity (spirometric) [grouped]

| anamnesis.copd_severity | N | % |
|-------------------------------------------------|----|----|
| COPD degree of severity (spirometric) [grouped] | IN | 70 |
| 1/2 | | |
| 3/4 | | |
| No preliminary examination result | | |
| Missing | | |
| Number of patients in Treated Set | | |

#### Table 15.1.4 9: mMRC Questionnaire

| mmrc.activity | N | % |
|--------------------|----|----|
| mMRC Questionnaire | IN | /0 |
| Grade 0 | | |
| Grade 1 | | |
| Grade 2 | | |
| Grade 3 | | |
| Grade 4 | | |

Final 3.0, 12.03.2019 8 / 53

| mmrc.activity | N | % |
|-----------------------------------|----|----|
| mMRC Questionnaire | IN | 70 |
| Missing | | |
| Number of patients in Treated Set | | |

Table 15.1.4 10: Treated Set- Exacerbations and hospitalizations due to excerbations in the last 12 months

| Exacerbations and hospitalizations due to | Number<br>of | Number of exa- | Mean | SD | Mean SD | SD Min | Median | Max | Nmiss | Patien<br>eve | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| excerbations in the last 12 months | patients | cerbations | | | | | | | | Z | % |
| anamnesis.exacerbation | | | | | | | | | | | |
| Number of exacerbations | | | | | | | | | | | |
| anamnesis.exacerbation_<br>hospital | | | | | | | | | | | |
| Number of hospitalizations due to excerbations | | | | | | | | | | | |

Table 15.1.4 11: Treated Set- Exacerbations and hospitalizations due to excerbations in the last 12 months, categorical

| anamnesis.exac | Hos | pitaliza | Number of patients in | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Exacerbations- Overview | | 0 | | | 1 2 | | 2 | | | Treated Set | |
| Exacerbation | is- Overview | N | % | N | % | N | % | N | N % N | | % |
| | 0 | | | | | | | | | | |
| Exacerbations in | 1 | | | | | | | | | | |
| the last 12<br>months | 2 | | | | | | | | | | |
| Number of patients in Treated Set | | | | | | | | | | | 100.0 |

Table 15.1.4 12: Treated Set- COPD degree of severity (GOLD group)

| COPD degree of severity (GOLD group) | N | % |
|--------------------------------------|---|---|
| A | | |
| В | | |
| С | | |
| D | | |
| Missing | | |
| Number of patients in Treated Set | | |

Final 3.0, 12.03.2019 9 / 53

Table 15.1.4 13: Treated Set- COPD degree of severity (GOLD group) [grouped]

| COPD degree of severity (GOLD group) [grouped] | N | % |
|------------------------------------------------|---|---|
| A/B | | |
| C/D | | |
| Missing | | |
| Number of patients in Treated Set | | |

Table 15.1.4 14: Treated Set- COPD degree of severity (GOLD group) - Distribution

| XXXXXXXXX | *************************************** | ŀ | 4 | | В | | С | | D | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|
| GOL | D stadium- Distribution | Ν | % | Ν | % | Z | % | Ν | % | Ν | % |
| Symptoms | Exacerbations | | | | | | | | | | |
| 0-1 | 0-1 | | | | | | | | | | |
| 0-1 | >=2 | | | | | | | | | | |
| 2-4 | 0-1 | | | | | | | | | | |
| 2-4 | >=2 | | | | | | | | | | |
| Number of pation | ents in Treated Set | | | | | | | | | | |

Table 15.1.4 15: Treated Set- COPD degree of severity (GOLD group) - Smoking

| COLD stadium Smaking | Α | | В | | С | | D | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|
| GOLD stadium- Smoking | Ν | % | Z | % | Ν | % | Z | % | Z | % |
| Smoker | | | | | | | | | | |
| Ex-smoker | | | | | | | | | | |
| Non-smoker | | | | | | | | | | |
| Missing | | | | | | | | | | |
| Number of patients in Treated Set | | | | | | | | | | |

Table 15.1.4 16: Treated Set- COPD degree of severity (GOLD group) - ICS at baseline

| GOLD stadium- ICS at baseline | Α | | В | | С | | D | | Missing | |
|---|---|---|---|---|---|---|---|---|---|---|
| GOLD stadium- ics at baseline | N | % | Ζ | % | Ν | % | Ν | % | Ν | % |
| No baseline ICS | | | | | | | | | | |
| ICS only at baseline | | | | | | | | | | |
| LABA+ICS at baseline | | | | | | | | | | |
| Missing | | | | | | | | | | |
| Number of patients in Treated Set | | | | | | | | | | |

Table 15.1.4 17: Treated Set- Patients with concomitant diseases

| anamnesis.disease | N | % |
|------------------------------------|----|----|
| Patients with concomitant diseases | IN | 70 |
| No | | |
| Yes | | |
| Missing | | |
| Number of patients in Treated Set | | |

Final 3.0, 12.03.2019 10 / 53

Table 15.1.4 18: Treated Set- Concomitant diseases (multiple answers possible)

| | | zases (muni |
|-----------------------------------|---|-------------|
| Concomitant diseases | N | % |
| anamnesis.disease_allergic | | |
| Allergic | | |
| anamnesis.disease_gastro | | |
| Gastrointestinal/Hepatobiliary | | |
| anamnesis.disease_pulmo | | |
| Pulmonary (except COPD) | | |
| anamnesis.disease_reproductive | | |
| Reproductive | | |
| anamnesis.disease_renal | | |
| Renal/Urogenital | | |
| anamnesis.disease_psychic | | |
| Psychiatric | | |
| anamnesis.disease_neuro | | |
| Neurologic | | |
| anamnesis.disease_cardiac | | |
| Cardial | | |
| anamnesis.disease_vascular | | |
| Vascular | | |
| anamnesis.disease_metabolic | | |
| Metabolic/Endocrine | | |
| anamnesis.disease_muscular | | |
| Muscular-skeletal/Dermatological | | |
| anamnesis.disease_other | | |
| Other | | |
| Number of patients in Treated Set | | |

Table 15.1.4 19: Treated Set- Concomitant diseases- Gastrointestinal/Hepatobiliary (multiple answers possible)

| Gastrointestinal/Hepatobiliary disease | N | % |
|-------------------------------------------------------|---|---|
| anamnesis.disease_gastro_gerd | | |
| Gastro-esophageal reflux disease (GERD) | | |
| anamnesis.disease_gastro_other | | |
| Other | | |
| Patients with gastrointestinal/hepatobiliary diseases | | |
| Number of patients in Treated Set | | |

Final 3.0, 12.03.2019 11 / 53

Table 15.1.4 20: Treated Set- Concomitant diseases- Pulmonary (except COPD) (multiple answers possible)

| Pulmonary (except COPD) | N | % |
|-----------------------------------|---|---|
| anamnesis.disease_pulmo_cancer | | |
| Lung cancer | | |
| anamnesis.disease_pulmo_other | | |
| Other | | |
| Patients with pulmonary diseases | | |
| Number of patients in Treated Set | | |

Table 15.1.4 21: Treated Set- Concomitant diseases- Metabolic/Endocrine (multiple answers possible)

| Metabolic/Endocrine | N | % |
|--------------------------------------------|---|---|
| anamnesis.disease_metabolic_dia | | |
| Diabetes mellitus | | |
| anamnesis.disease_metabolic_oth | | |
| Other | | |
| Patients with metabolic/endocrine diseases | | |
| Number of patients in Treated Set | | |

Table 15.1.4 22: Treated Set- Concomitant diseases- Muscular-skeletal/ Dermatological (multiple answers possible)

| · | |
|----------------------------------------------------------|---|
| Muscular-skeletal/Dermatological | % |
| anamnesis.disease_muscular_osteo | |
| Osteoporosis | |
| anamnesis.disease_muscular_other | |
| Other | |
| Patients with muscular-skeletal/ dermatological diseases | |
| Number of patients in Treated Set | |

Table 15.1.4 23: Treated Set- Smoking

| anamnesis.smoker | N | % |
|-----------------------------------|----|----|
| Smoking | IN | 70 |
| Smoker | | |
| Ex-smoker | | |
| Non-smoker | | |
| Missing | | |
| Number of patients in Treated Set | | |

Final 3.0, 12.03.2019 12 / 53

Table 15.1.4 24: Treated Set- Smoking- Pack-years

| anamnesis.smoker_pack_years | N | Mean | SD | Min | Median | Max | Nmiss |
|-----------------------------|---|------|----|-----|--------|-----|-------|
| Pack-years | | | | | | | |

Table 15.1.4 25: Treated Set- Patients with concomitant medication (except respiratory therapeutics)

| anamnesis.medication | N | % |
|-----------------------------------|----|----|
| Concomitant medication | IN | 70 |
| No | | |
| Yes | | |
| Missing | | |
| Number of patients in Treated Set | | |

Table 15.1.4 26: Treated Set- Diseases treated with concomitant medication (except respiratory therapeutics)- (multiple answers possible)

| anamnesis_medication.disease | N | % |
|---|---|---|
| Concomitant medication- Disease treated | IN | /0 |
| Allergic | | |
| Gastrointestinal/Hepatobiliary- Gastro esophageal reflux disease (GERD) | | |
| Gastrointestinal/Hepatobiliary- Other | | |
| Pulmonary (except COPD)- Lung cancer | | |
| Pulmonary (except COPD)- Other | | |
| Reproductive | | |
| Renal/Urogenital | | |
| Psychiatric | | |
| Neurologic | | |
| Cardial | | |
| Vascular | | |
| Metabolic/Endocrine- Diabetes mellitus | | |
| Metabolic/Endocrine- Other | | |
| Muscular-skeletal/Dermatological- Osteoporosis | | |
| Muscular-skeletal/Dermatological- Other | | |
| Other | | |
| Number of patients in Treated Set | | |

Table 15.1.4 27: Treated Set- Concomitant medication (except respiratory therapeutics)-Continuation or new prescription (multiple answers possible)

| anamnesis_medication.type | N | % |
|----------------------------------------------------------|----|----|
| Concomitant medication- Continuation or new prescription | IN | /0 |
| Continuation | | |
| New prescription | | |
| Missing | | |
| Number of patients in Treated Set | | |

Final 3.0, 12.03.2019 13 / 53

Table 15.1.4 28: Treated Set- Spiolto<sup>®</sup> Respimat<sup>®</sup> - Patient trained to use inhaler

| anamnesis.spiolto_training | N | % |
|-----------------------------------|----|----|
| Patient trained to use inhaler | IN | 70 |
| No | | |
| Yes | | |
| Missing | | |
| Number of patients in Treated Set | | |

Table 15.1.4 29: Treated Set- Treatment with past COPD therapies (6 weeks prior to start of study treatment) according to mMRC value

| | | mMRC value | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| anamnesis.respiratory | Grade 0 | | Grade 1 | | Grade 2 | | Grade 3 | | Grade 4 | | Total | |
| Treatment with past COPD therapies | Ν | % | N | % | N | % | Ν | % | Ν | % | N | % |
| No | | | | | | | | | | | | |
| Yes | | | | | | | | | | | | |
| Missing | | | | | | | | | | | | |
| Number of patients in Treated Set | | | | | | | | | | | | |

Table 15.1.4 30: Treated Set- Treatment with past COPD therapies (6 weeks prior to start of study treatment)- Respiratory therapeutics (multiple answers possible)

| anamnesis_resp.therapy/anamnesis_resp_prescribe | With | drawn | N | ew | Conti | nued | Miss | sing |
|---|---|---|---|---|---|---|---|---|
| Treatment with past COPD therapies- Therapeutics | N | % | N | % | N | % | N | % |
| Short-acting β <sub>2</sub> -Agonist | | | | | | | | |
| Long-acting β <sub>2</sub> -Agonist | | | | | | | | |
| Short-acting anticholinergic | | | | | | | | |
| Long-acting anticholinergic | | | | | | | | |
| Long-acting anticholinergic and long-acting $\beta_2$ -Agonist in a fixed combination | | | | | | | | |
| Short-acting anticholinergic and short-acting β <sub>2</sub> -Agonist in a fixed combination | | | | | | | | |
| Long-acting $\beta_2$ -Agonist and inhaled corticosteroid in a fixed combination | | | | | | | | |
| Inhaled corticosteroid | | | | | | | | |
| Systemic corticosteroid | | | | | | | | |
| Theophylline | | | | | | | | |
| Roflumilast (Daxas <sup>®</sup> ) | | | | | | | | |
| Other | | | | | | | | |
| Missing | | | | | | | | |
| Number of patients in Treated Set | | | | | | | | |

Final 3.0, 12.03.2019 14 / 53

#### Visit 2 (after approx. 6 weeks of therapy)

Table 15.1.4 31: Treated Set- Therapy with Spiolto® Respimat® carried out regularly

| visit.spiolto_regular | N | % |
|-------------------------------------------------------|----|----|
| Therapy with Spiolto® Respimat® carried out regularly | IN | 70 |
| No | | |
| Yes | | |
| Missing | | |
| Number of patients in Treated Set with visit 2 | | |

Table 15.1.4 32: Treated Set- Reason for therapy with Spiolto<sup>®</sup> Respimat<sup>®</sup> carried out irregularly

| visit.spiolto_regular_reason | N | % |
|---------------------------------------------|----|----|
| Reason for irregular treatment | IN | 70 |
| Adverse event | | |
| Serious adverse event | | |
| Patient's wish | | |
| Other | | |
| Missing | | |
| Number of patients with irregular treatment | | |

Table 15.1.4 33: Treated Set- Changes of treatment with other COPD related therapies besides Spiolto<sup>®</sup> Respimat<sup>®</sup> since visit 1 [i.e. new therapy introduced or existing baseline therapy discontinued\*]

| visit.further_resp | N | % |
|--------------------------------------------------------|----|----|
| Changes of treatment with other COPD related therapies | IN | 70 |
| No | | |
| Yes | | |
| Missing | | |
| Number of patients in Treated Set with visit 2 | | _ |

<sup>\*</sup>New therapy: New therapy in addition to already existing baseline therapies besides Spiolto® Respimat®

Table 15.1.4 34: Treated Set- Changes of treatment with other COPD related therapies besides Spiolto<sup>®</sup> Respimat<sup>®</sup> since visit 1- Affected respiratory therapeutics (multiple answers possible)

| | visit_resp.therapeutic | N | % |
|---|---|---|---|
| Changes | of treatment with other COPD related therapies- Affected therapeutics | 1 | 70 |
| | Short-acting β <sub>2</sub> -Agonist | | |
| | Long-acting β <sub>2</sub> -Agonist | | |
| New therapy in | Short-acting anticholinergic | | |
| addition to already existing baseline | Long-acting anticholinergic | | |
| therapies besides | Long-acting anticholinergic and long-acting $\beta_2$ -Agonist in a fixed combination | | |
| Spiolto <sup>®</sup> Respimat <sup>®</sup> introduced after | Short-acting anticholinergic and short-acting $\beta_2$ -Agonist in a fixed combination | | |
| visit 1 | Long-acting β <sub>2</sub> -Agonist and inhaled corticosteroid in a fixed combination | | |
| | Inhaled corticosteroid | | |
| | Systemic corticosteroid | | |

Final 3.0, 12.03.2019 15 / 53

| ****** | visit_resp.therapeutic | N | % |
|---|---|---|---|
| Changes | of treatment with other COPD related therapies- Affected therapeutics | | /0 |
| | Theophylline | | |
| | Roflumilast (Daxas <sup>®</sup> ) | | |
| | Other | | |
| | Number of patients in Treated Set with visit 2 | | |
| | Short-acting β <sub>2</sub> -Agonist | | |
| | Long-acting β <sub>2</sub> -Agonist | | |
| | Short-acting anticholinergic | | |
| | Long-acting anticholinergic | | |
| | Long-acting anticholinergic and long-acting β <sub>2</sub> -Agonist in a fixed combination | | |
| Components of existing baseline | Short-acting anticholinergic and short-acting $\beta_2$ -Agonist in a fixed combination | | |
| therapy at visit 1 | Long-acting β <sub>2</sub> -Agonist and inhaled corticosteroid in a fixed combination | | |
| discontinued since then | Inhaled corticosteroid | | |
| unon | Systemic corticosteroid | | |
| | Theophylline | | |
| | Roflumilast (Daxas <sup>®</sup> ) | | |
| | Other | | |
| | Number of patients in Treated Set with visit 2 | | |

Table 15.1.4 35: Treated Set- Changes of concomitant diseases since visit 1 [i.e. new diagnosis or now-defunct diagnosis]

| visit.disease | N | % |
|------------------------------------------------|----|----|
| Changes of concomitant diseases | IN | 70 |
| No | | |
| Yes | | |
| Missing | | |
| Number of patients in Treated Set with visit 2 | | |

Table 15.1.4 36: Treated Set- Changes of concomitant diseases- Diseases (multiple answers possible)

| visit_disease.disease | | N | % |
|---|---|---|---|
| | Changes of concomitant diseases- Diseases | IN | 70 |
| | Allergic | | |
| | Gastrointestinal/Hepatobiliary- Gastro esophageal reflux disease (GERD) | | |
| | Gastrointestinal/Hepatobiliary- Other | | |
| A new | Pulmonary (except COPD)- Lung cancer | | |
| diagnosis after | Pulmonary (except COPD)- Other | | |
| visit 1 | Reproductive | | |
| | Renal/Urogenital | | |
| | Psychiatric | | |
| | Neurologic | | |

Final 3.0, 12.03.2019 16 / 53

| | visit_disease.disease | N | % |
|---|---|---|---|
| | Changes of concomitant diseases- Diseases | IN | /0 |
| | Cardial | | |
| | Vascular | | |
| | Metabolic/Endocrine- Diabetes mellitus | | |
| | Metabolic/Endocrine- Other | | |
| | Muscular-skeletal/Dermatological- Osteoporosis | | |
| | Muscular-skeletal/Dermatological- Other | | |
| | Other | | |
| | Number of patients in Treated Set with visit 2 | | |
| | Allergic | | |
| | Gastrointestinal/Hepatobiliary- Gastro esophageal reflux disease (GERD) | | |
| | Gastrointestinal/Hepatobiliary- Other | | |
| | Pulmonary (except COPD)- Lung cancer | | |
| | Pulmonary (except COPD)- Other | | |
| | Reproductive | | |
| | Renal/Urogenital | | |
| Existing | Psychiatric | | |
| diagnosis at visit 1 now- | Neurologic | | |
| defunct | Cardial | | |
| | Vascular | | |
| | Metabolic/Endocrine- Diabetes mellitus | | |
| | Metabolic/Endocrine- Other | | |
| | Muscular-skeletal/Dermatological- Osteoporosis | | |
| | Muscular-skeletal/Dermatological- Other | | |
| | Other | | |
| | Number of patients in Treated Set with visit 2 | | |

Table 15.1.4 37: Treated Set- Changes of concomitant medication since visit 1 [i.e. new medication introduced or existing medication discontinued]

| visit.medication | N | % |
|------------------------------------------------|----|----|
| Changes of concomitant medication | IN | 70 |
| No | | |
| Yes | | |
| Missing | | |
| Number of patients in Treated Set with visit 2 | | |

Final 3.0, 12.03.2019 17 / 53

Table 15.1.4 38: Treated Set- Changes of concomitant medication- Disease treated

| ****** | visit_medication.disease | N | % |
|---|---|---|---|
| | Changes of concomitant medication- Disease treated | IN | 70 |
| | Allergic | | |
| | Gastrointestinal/Hepatobiliary- Gastro esophageal reflux disease (GERD) | | |
| | Gastrointestinal/Hepatobiliary- Other | | |
| | Pulmonary (except COPD)- Lung cancer | | |
| | Pulmonary (except COPD)- Other | | |
| | Reproductive | | |
| | Renal/Urogenital | | |
| New | Psychiatric | | |
| medication | Neurologic | | |
| after visit 1 | Cardial | | |
| | Vascular | | |
| | Metabolic/Endocrine- Diabetes mellitus | | |
| | Metabolic/Endocrine- Other | | |
| | Muscular-skeletal/Dermatological- Osteoporosis | | |
| | Muscular-skeletal/Dermatological- Other | | |
| | Other | | |
| | Number of patients in Treated Set with visit 2 | | |
| | Allergic | | |
| | Gastrointestinal/Hepatobiliary- Gastro esophageal reflux disease (GERD) | | |
| | Gastrointestinal/Hepatobiliary- Other | | |
| | Pulmonary (except COPD)- Lung cancer | | |
| | Pulmonary (except COPD)- Other | | |
| | Reproductive | | |
| | Renal/Urogenital | | |
| Existing medication | Psychiatric | | |
| at visit 1 | Neurologic | | |
| discontinued since then | Cardial | | |
| Silice then | Vascular | | |
| | Metabolic/Endocrine- Diabetes mellitus | | |
| | Metabolic/Endocrine- Other | | |
| | Muscular-skeletal/Dermatological- Osteoporosis | | |
| | Muscular-skeletal/Dermatological- Other | | |
| | Other | | |
| | Number of patients in Treated Set with visit 2 | | |

Final 3.0, 12.03.2019 18 / 53

Table 15.1.4 39: Treated Set- Smokers at baseline- Current status (smoking status at visit 2)

| visit.smoker | N | % |
|-----------------------------------------------------------|---|---|
| Smoker at baseline- Current status | | |
| Patient still smokes | | |
| Patient stopped smoking | | |
| Missing | | |
| Number of smokers at baseline in Treated Set with visit 2 | | |

Table 15.1.4 40: Treated Set- Pregnancy during treatment

| visit.pregnancy | N | % |
|-------------------------------------------------------|----|----|
| Pregnancy during treatment | IN | 70 |
| No | | |
| Yes | | |
| Number of female patients in Treated Set with visit 2 | | |

Final 3.0, 12.03.2019

#### 2.2.1.1.4 15.2. Efficacy evaluation

#### **Primary endpoints**

Table 15.2.1 1: Full Analysis Set- Total CCQ score- Share of patients with therapeutic success after 6 weeks (approximately), defined as 0.4-point decrease of total CCQ score between baseline and week 6 (approximately)

| CCQ Share of patients with therapeutic success | N | %* | CI 95% |
|------------------------------------------------|---|----|--------|
| Therapy successful | | | |
| Therapy not successful | | | |
| Missing | | | |
| Total | | | |

<sup>\*</sup>percentage is based on the total number of patients, irrespective of the availability of the CCQ score

Table 15.2.1 2: Full Analysis Set- CCQ score

| <u> </u> | CCQ<br>CCQ score | N | Mean | CI 95% | Std | Min | Median | Max | Nmiss |
|---|---|---|---|---|---|---|---|---|---|
| | Symptom | | | | | | | | |
| Baseline | Functional state (CCQ-4) | | | | | | | | |
| (Visit 1) | Mental state | | | | | | | | |
| | Total CCQ score | | | | | | | | |
| | Symptom | | | | | | | | |
| Week 6<br>(appr.)<br>(Visit 2) | Functional state (CCQ-4) | | | | | | | | |
| | Mental state | | | | | | | | |
| | Total CCQ score | | | | | | | | |

#### Secondary endpoints

Table 15.2.1 3: Full Analysis Set- Absolut change of CCQ score between baseline and week 6 (approximately)

| CCQ CCQ score- Change between baseline and Week 6 (approximately) | Ν | Mean | CI 95% | Std | Min | Median | Max | Nmiss |
|---|---|---|---|---|---|---|---|---|
| Symptom | | | | | | | | |
| Functional state (CCQ-4) | | | | | | | | |
| Mental state | | | | | | | | |
| Total CCQ score | | | | | | | | |

Final 3.0, 12.03.2019 20 / 53

Table 15.2.1 4: Full Analysis Set- General condition of the patient evaluated by the physician (PGE- score)

| General condition of patient (PGE score)* | | % |
|-------------------------------------------|------------------------|---|
| anamnesis.general_condition 1 | | |
| | 2 | |
| | 3 | |
| | 4 | |
| | 5 | |
| Baseline (Visit 1) | 6 | |
| | 7 | |
| | 8 | |
| | Missing | |
| | Number of patients | |
| visit.general_condition | 1 | |
| | 2 | |
| | 3 | |
| | 4 | |
| | 5 | |
| Week 6 (approximately) (Visit 2) | 6 | |
| | 7 | |
| | 8 | |
| | Missing/Not applicable | |
| | Number of patients | |

<sup>\*</sup>poor=1-2, satisfactory=3-4, good=5-6, excellent=7-8

Table 15.2.1 5: Full Analysis Set- Patient satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup>

| Patient satisfaction | | N | % |
|---|---|---|---|
| visit.satisfaction_spiolto | Very satisfied | | |
| Patient overall satisfaction with Spiolto <sup>®</sup> Respimat <sup>®</sup> treatment | Satisfied | | |
| | Rather satisfied | | |
| | Neither satisfied nor dissatisfied | | |
| | Rather dissatisfied | | |
| | Dissatisfied | | |
| opiolo respinar acamen | Very dissatisfied | | |
| | Not answered | | |
| | Missing | | |
| | Total | | |
| visit.satisfaction_inhalator | Very satisfied | | |
| Patient satisfaction with inhaling from | Satisfied | | |
| the Respimat <sup>®</sup> device | Rather satisfied | | |

Final 3.0, 12.03.2019 21 / 53

| Patient satisfaction | | % |
|---|---|---|
| | Neither satisfied nor dissatisfied | |
| | Rather dissatisfied | |
| | Dissatisfied | |
| | Very dissatisfied | |
| | Not answered | |
| | Missing | |
| Total | | |
| visit.satisfaction_handling Very satisfied | | |
| | Satisfied | |
| | Rather satisfied | |
| | Neither satisfied nor dissatisfied | |
| | Rather dissatisfied | |
| Patient satisfaction with handling of the Respimat® inhalation device | Dissatisfied | |
| the respinal inhalation device | Very dissatisfied | |
| | Not answered | |
| | Missing | |
| | Total | |

Table 15.2.1 6: Full Analysis Set- Patient's willingness to continue Spiolto® Respimat®

| visit.spiolto_continued | N | % |
|---------------------------------|----|----|
| Willing to continue treatment | IN | 70 |
| Yes | | |
| No | | |
| Missing | | |
| Number of patients with visit 2 | | |

Table 15.2.1 7: Full Analysis Set- Reason for discontinuation of Spiolto® Respimat®

| visit.spiolto_spiolto_reason | N | % |
|--------------------------------------|----|----|
| Reason for treatment discontinuation | IN | /0 |
| Adverse event | | |
| Serious adverse event | | |
| Patient's wish | | |
| Withdrawal of informed consent | | |
| Lost to follow-up | | |
| Patient's death | | |
| Other | | |
| Missing | | |
| Number of patients with visit 2 | | |

Final 3.0, 12.03.2019 22 / 53

## 2.2.1.1.5 15.3. Safety analysis

#### Extent of exposure

Table 15.3.1 1: Treated Set- Time between start of treatment and end of observation/discontinuation [weeks]

| anamnesis.spiolto_date; visit.date; visit.spiolto_last_date | N | Mean | Std | Min | Median | Max | Nmiss |
|---|---|---|---|---|---|---|---|
| Time between start of treatment and end of observation/discontinuation | | | | | | | |

Table 15.3.1 2: Treated Set- Survival status

| sae.therapy; visit.done_reason | N | % |
|--------------------------------|----|----|
| Survival status | IN | 70 |
| Patient died | | |
| Patient alive | | |
| No. of patients in Treated Set | | |

## Safety

Table 15.3.2 1: Treated Set- Adverse events overall summary

| | N (%) |
|---|---|
| Number of patients | xx (100.0) |
| Patients with investigator defined drug-related AE {sae.spiolto_causality} | xx (yy.y) |
| Patients with investigator defined drug-related AE leading to discontinuation of trial drug {sae.spiolto_action_taken} | xx (yy.y) |
| Patients with serious AE {sae.sae} | xx (yy.y) |
| Fatal {sae.criteria_fatal} | xx (yy.y) |
| Life threatening {sae.criteria_life_theratening} | xx (yy.y) |
| Persistant or significant disability/incapacity {sae.criteria_disability} | xx (yy.y) |
| Hospitalization {sae.criteria_hospital} | xx (yy.y) |
| Prolongation of hospitalization necessary {sae.criteria_prolonged} | xx (yy.y) |
| Congenital anomaly/birth defect {sae.criteria_congenital} | xx (yy.y) |
| Other important medical event {sae.criteria_other} | xx (yy.y) |
| Patients with serious AE leading to discontinuation {sae.sae} {sae.spiolto_action_taken} | xx (yy.y) |
| Patients with serious drug-related AE {sae.sae} {sae.spiolto_causality} | xx (yy.y) |

### Drug-related adverse events (Drug-related AE)

Table 15.3.2 2: Treated Set- Drug-related AE according to MedDRA-SOC and PT (event based)

| Sac | :.nci | N | % |
|----------------|-------|----|---|
| Drug-related A | IN | 70 | |
| | PT1 | | |
| SOC1 | PT2 | | |
| | PT1 | | |
| SOC2 | PT2 | | |

Final 3.0, 12.03.2019 23 / 53

| sae | sae.nci | | % |
|-----------------|---------|----|---|
| Drug-related Al | N | /0 | |
| | PT1 | | |
| | PT2 | | |
| Total | | | |

Table 15.3.2 3: Treated Set- Drug-related AE by MedDRA system organ class and preferred term- Maximum NCI grade per patient

| **** | sae.nci | Gra | de 1 | Gra | de 2 | Gra | de 3 | Gra | de 4 | Gra | de 5 | То | tal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | ited AE-Maximum<br>le per patient | Ν | % | N | % | N | % | N | % | N | % | N | % |
| Any SOC | | | | | | | | | | | | | |
| | PT1 | | | | | | | | | | | | |
| SOC1 | PT2 | | | | | | | | | | | | |
| | PT1 | | | | | | | | | | | | |
| SOC2 | PT2 | | | | | | | | | | | | |
| | PT1 | | | | | | | | | | | | |
| | PT2 | | | | | | | | | | | | |
| No. of patie | ents in Treated Set | | | | | | | | | | | | |

Table 15.3.2 4: Treated Set- Number of patients with drug-related AE occurring with share in preferred term greater than 5% by primary system organ class and preferred term

| | N (%) |
|---|---|
| Total with drug-related AE occurring with share in preferred term greater than 5% | xx (100.0) |
| Primary SOC {sae.nci} | xx (yy.y) |
| Preferred term | xx (yy.y) |
| | xx (yy.y) |

Table 15.3.2 5: Treated Set- Drug-related AE- Worst outcome per patient

| sae.outcome | N | % |
|----------------------------------|----|-----|
| Drug-related AE- Worst outcome | IN | -/0 |
| Recovered/Resolved | | |
| Not yet recovered/resolved | | |
| Recovered/resolved with sequelae | | |
| Fatal | | |
| Unknown | | |
| No drug-related AE | | |
| No. of patients in Treated Set | | |

Order: From best to worst: Recovered/resolved; Recovered/resolved with sequelae; Not recovered/Not resolved; Unknown; Fatal

Final 3.0, 12.03.2019 24 / 53

Table 15.3.2 6: Treated Set- Drug-related AE- Patients with at least one drug-related AE for which therapy was required

| sae.therapy | N | % |
|-----------------------------------|----|----|
| Drug-related AE- Therapy required | IN | 70 |
| No | | |
| Yes | | |
| Missing | | |
| No drug-related AE | | |
| No. of patients in Treated Set | | |

Table 15.3.2 7: Treated Set- Drug-related AE- Patient pregnant at AE

| sae.pregnancy | N | % |
|---------------------------|----|----|
| Drug-related AE- Pregnant | IN | 70 |
| No | | |
| Yes | | |
| Not applicable | | |
| Missing | | |
| Total | | |

Table 15.3.2 8: Treated Set- Drug-related AE- Week of pregnancy

| sae.pregnancy_week | N | Mean | SD | Min | Median | Max | Nmiss |
|---|---|---|---|---|---|---|---|
| Drug-related AE- Week of pregnancy | | | | | | | |

Table 15.3.2 9: Treated Set- Drug-related AE- Action taken concerning therapy (patient based; multiple answers possible)

| sae.nci; sae.spiolto_action_taken | N | % |
|--------------------------------------|----|----|
| Drug-related AE- Action taken | IN | 70 |
| Continued | | |
| Reduced | | |
| Stopped | | |
| Increased | | |
| Missing | | |
| No. of patients with drug-related AE | | |

Table 15.3.2 10: Treated Set- Drug-related AE leading to treatment discontinuation by MedDRA system organ class and preferred term

| ***** | sae.nci | N | % |
|----------------|---------|----|---|
| Drug-related A | IN | /0 | |
| Any SOC | | | |
| | PT1 | | |
| SOC1 | PT2 | | |
| 5002 | PT1 | | |
| SOC2 | PT2 | | |

Final 3.0, 12.03.2019 25 / 53

| sae.nci | | N | % |
|---|---|---|---|
| Drug-related AE leading to discontinuation (patient based) | | | /0 |
| | :: | | |
| | PT1 | | |
| | PT2 | | |
| No. of patients in | Treated Set | | |

Table 15.3.2 11: Treated Set- Drug-related AE- Improvement after stop of therapy (patient based; multiple answers possible)

| sae.spiolto_action_taken_stop | N | % |
|-------------------------------------------------------------------|----|----|
| Drug-related AE- Improvement after stop | IN | 70 |
| No | | |
| Yes | | |
| Missing | | |
| No. of patients with stop of treatment because of drug-related AE | | |

Table 15.3.2 12: Treated Set- Drug-related AE- Re-exposition done for at least one event

| sae.spiolto_action_taken_expo | N | % |
|-------------------------------------------------------------------|----|----|
| Drug-related AE- Re-exposition | ., | 70 |
| No | | |
| Yes | | |
| Not applicable | | |
| Missing | | |
| No. of patients with stop of treatment because of drug-related AE | | |

Table 15.3.2 13: Treated Set- Drug-related AE- Recurrence of at least one TEAE after reexposition

| sae.spiolto_action_taken_again | N | % |
|-------------------------------------------------|---|---|
| Drug-related AE- Recurrence after re-exposition | | |
| No | | |
| Yes | | |
| Missing | | |
| No. of patients with re-exposition | | |

Table 15.3.2 14: Treated Set-Incorrect administration of medication (multiple answers possible)

| Incorrect administration of medication | N | % |
|----------------------------------------|---|---|
| sae.application_abuse | | |
| Abuse/Incorrect use | | |
| sae.application_medication_error | | |
| Medication error | | |
| sae.application_overdose | | |

Final 3.0, 12.03.2019 26 / 53

| Incorrect administration of medication | N | % |
|-----------------------------------------|---|---|
| Overdosing | | |
| sae.application_other | | |
| Other | | |
| Patients with incorrect administration | | |
| Number of patients with drug-related AE | | |

### Serious AE

Table 15.3.2 15: Treated Set- Serious AE according to MedDRA-SOC and PT (event based)

| sae.nci; | sae.sae | NI | % |
|--------------|--------------|----|----|
| Serious AE ( | event based) | N | 70 |
| | PT1 | | |
| SOC1 | PT2 | | |
| | PT1 | | |
| SOC2 | PT2 | | |
| | PT1 | | |
| PT2 | | | |
| Total | | | |

Table 15.3.2 16: Treated Set- Serious AE- Reason for seriousness (patient based; multiple answers possible)

| Reason for serious AE | N | % |
|------------------------------------------------|---|---|
| sae.criteria_fatal | | |
| Fatal | | |
| sae.criteria_life_threatening | | |
| Life threatening | | |
| sae.criteria_disability | | |
| Sustained or significant disability/incapacity | | |
| sae.criteria.hospital | | |
| Hospitalization required | | |
| sae.criteria_prolonged | | |
| Hospitalization extended | | |
| sae.criteria_congenital | | |
| Congenital anomaly | | |
| sae.criteria_other | | |
| Otherwise medically significant | | |
| Number of patients with serious AE | | |

Final 3.0, 12.03.2019 27 / 53

Table 15.3.2 17: Treated Set- Serious AE by MedDRA system organ class and preferred term-Maximum NCI grade per patient

| XXXXXX | sae.nci | Gra | de 1 | Gra | de 2 | Gra | de 3 | Gra | de 4 | Gra | de 5 | То | tal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Serious A | AE- Maximum grade per patient | N | % | Ν | % | N | % | N | % | N | % | N | % |
| Any SOC | | | | | | | | | | | | | |
| | PT1 | | | | | | | | | | | | |
| SOC1 | PT2 | | | | | | | | | | | | |
| | PT1 | | | | | | | | | | | | |
| SOC2 | PT2 | | | | | | | | | | | | |
| | PT1 | | | | | | | | | | | | |
| | PT2 | | | | | | | | | | | | |
| No. of patie | ents in Treated Set | | | | | | | | | | | | |

Table 15.3.2 18: Treated Set- Serious AE- Worst outcome per patient

| sae.outcome; sae.sae | N | % |
|----------------------------------|----|----|
| Serious AE- Outcome | IN | 70 |
| Recovered/Resolved | | |
| Not yet recovered/resolved | | |
| Recovered/resolved with sequelae | | |
| Fatal | | |
| Unknown | | |
| No serious AE | | |
| No. of patients in Treated Set | | |

Order: From best to worst: Recovered/resolved; Recovered/resolved with sequelae; Not recovered/Not resolved; Unknown; Fatal

Table 15.3.2 19: Treated Set- Serious AE- Action taken concerning treatment (patient based; multiple answers possible)

| sae.nci; sae.spiolto_action_taken | N | % |
|-----------------------------------|----|----|
| Serious AE- Action taken | IN | 70 |
| Continued | | |
| Reduced | | |
| Stopped | | |
| Increased | | |
| Missing | | |
| No. of patients with serious AE | | |

Final 3.0, 12.03.2019 28 / 53

Table 15.3.2 20: Treated Set- Serious AE leading to treatment discontinuation by MedDRA system organ class and preferred term

| ******* | sae.nci | N | % |
|---|---|---|---|
| Serious AE lea | Serious AE leading to discontinuation (patient based) | | |
| Any SOC | | | |
| | PT1 | | |
| SOC1 | PT2 | | |
| | PT1 | | |
| SOC2 | PT2 | | |
| | PT1 | | |
| | PT2 | | |
| No. of patients in | Treated Set | | |

Table 15.3.2 21: Treated Set- Serious AE- Number of patients with at least one serious AE with causal relationship to treatment

| sae.causality | N | % |
|--------------------------|----|----|
| Serious AE- Relationship | IN | /0 |
| No | | |
| Yes | | |
| Missing | | |
| Total | | |

Table 15.3.2 22: Treated Set- Serious AE by relationship with Spiolto<sup>®</sup> Respimat<sup>®</sup> by MedDRA system organ class and preferred term

| sae.nci; sae.spiolto_causality | | Not related | | Rela | ated | Total | |
|---|---|---|---|---|---|---|---|
| Serious AE by relationship (patient based) | | N | % | N | % | N | % |
| Any SOC | | | | | | | |
| | PT1 | | | | | | |
| SOC1 | PT2 | | | | | | |
| | PT1 | | | | | | |
| SOC2 | PT2 | | | | | | |
| | PT1 | | | | | | |
| | PT2 | | | | | | |
| No. of patie | ents in Treated Set | | | | | | |

Final 3.0, 12.03.2019 29 / 53

#### 2.3 Sensitivity analysis I- Time between Visit 1 and Visit 2

#### Sensitivity analysis- Table 1: Full Analysis Set- Time between Visit 1 and Visit 2 [weeks]

| Anamnesis.date.; visit.date | Mean | Std | Min | Median | Max | Nmiss |
|---|---|---|---|---|---|---|
| Sensitivity analysis I- Time between Visit 1 and Visit 2 | | | | | | |

#### Sensitivity analysis- Table 2: Full Analysis Set- Time between Visit 1 and Visit 2 [categorical]

| Anamnesis.date.; visit.date |
|---|
| Sensitivity analysis I- Time between Visit 1 and Visit 2 [categorical] |
| < 4 weeks |
| 4-8 weeks |
| > 8 weeks |
| Patients in FAS |

Sensitivity analysis- Table 3: Analysis stratified by time between Visit 1 and Visit 2- Full Analysis Set- Total CCQ score- Share of patients with therapeutic success after 6 weeks (approximately)- defined as 0.4-point decrease of total CCQ score between baseline and week 6 (approximately)

| C | | | |
|-----------------------------------|------------------------|---|--------|
| Sensitivity analysis I- Share suc | N | % | CI 95% |
| | Therapy successful | | |
| < 4 weeks | Therapy not successful | | |
| ~ 4 WEEKS | Missing | | |
| | Total | | |
| | Therapy successful | | |
| 4-8 weeks | Therapy not successful | | |
| | Missing | | |
| | Total | | |
| | Therapy successful | | |
| > 8 weeks | Therapy not successful | | |
| > o weeks | Missing | | |
| | Total | | |
| | Therapy successful | | |
| Total | Therapy not successful | | |
| TUlai | Missing | | |
| | Total | | |

Sensitivity analysis- Table 4: Analysis stratified by time between Visit 1 and Visit 2- Full Analysis Set- Total CCQ score- Share of patients with therapeutic success-  $\chi^2$ -Test (Fisher's Exact test)

| Therapy success | p-Value |
|-------------------------------|---------|
| X²-Test (Fisher's Exact test) | |

Final 3.0, 12.03.2019 30 / 53

# Sensitivity analysis- Table 5: Analysis stratified by time between Visit 1 and Visit 2- Full Analysis Set- CCQ score

| XXXXXXX | ccq | XXXXXXX | N | Mean | CI | Std | Min | Median | Max | Nmiss |
|---|---|---|---|---|---|---|---|---|---|---|
| Sensitiv | Sensitivity analysis I- CCQ score | | IN | ivicari | 95% | Siu | IVIIII | Median | IVIAX | IVIIIISS |
| | | < 4 weeks | | | | | | | | |
| | Symptom | 4-8 weeks | | | | | | | | |
| | Symptom | > 8 weeks | | | | | | | | |
| | | Total | | | | | | | | |
| | | < 4 weeks | | | | | | | | |
| | Functional | 4-8 weeks | | | | | | | | |
| | state (CCQ-4) | > 8 weeks | | | | | | | | |
| Baseline<br>(Visit 1) | | Total | | | | | | | | |
| (VISIL I) | | < 4 weeks | | | | | | | | |
| | Montal atata | 4-8 weeks | | | | | | | | |
| | Mental state | > 8 weeks | | | | | | | | |
| | | Total | | | | | | | | |
| | Total CCQ<br>score | < 4 weeks | | | | | | | | |
| | | 4-8 weeks | | | | | | | | |
| | | > 8 weeks | | | | | | | | |
| | | Total | | | | | | | | |
| | | < 4 weeks | | | | | | | | |
| | C) mantama | 4-8 weeks | | | | | | | | |
| | Symptom | > 8 weeks | | | | | | | | |
| | | Total | | | | | | | | |
| | | < 4 weeks | | | | | | | | |
| | Functional | 4-8 weeks | | | | | | | | |
| | state (CCQ-4) | > 8 weeks | | | | | | | | |
| Week 6 | | Total | | | | | | | | |
| (appr.) (Visit<br>2) | | < 4 weeks | | | | | | | | |
| , | Montal atata | 4-8 weeks | | | | | | | | |
| | Mental state | > 8 weeks | | | | | | | | |
| | | Total | | | | | | | | |
| | | < 4 weeks | | | | | | | | |
| | Total CCQ | 4-8 weeks | | | | | | | | |
| | score | > 8 weeks | | | | | | | | |
| | | Total | | | | | | | | |

Final 3.0, 12.03.2019 31 / 53

### 2.4 Sensitivity analysis II- Non-estimated number of exacerbations\*

\*If the physician does not know the exact number of exacerbations he is allowed to give an estimate. In this analysis only those documentations are considered in which the physician knew the exact number, i.e. the number is not estimated (non-estimated).

# Sensitivity analysis- Table 6: Full Analysis Set- Patients with non-estimated number of exacerbations

| anamnesis.estimate | | |
|----------------------------------------------------------------|---|---|
| Sensitivity analysis II- Non-estimated number of exacerbations | N | % |
| No | | |
| Yes | | |
| Patients in FAS | | |

# Sensitivity analysis- Table 7: Full Analysis Set- Patients with non-estimated number of exacerbations- Exacerbations in the last 12 months

| anamnesis.exacerbation | of e | Number of exa- | Mean | SD | Min | Median | Max | Nmiss | Patients with event | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | cerbations | | | | | | | N | % |
| Sensitivity analysis II-<br>Exacerbations in the last 12<br>months | | | | | | | | | | |

# Sensitivity analysis- Table 8: Full Analysis Set- Patients with non-estimated number of exacerbations- Exacerbations in the last 12 months [categorical]

| anamnesis.exacerbation; | | |
|---|---|---|
| Sensitivity analysis II- Exacerbations in the last 12 months- Overview | N | % |
| No | | |
| Yes | | |
| Patients in FAS with non-estimated number of exacerbations | | |

# Sensitivity analysis- Table 9: Full Analysis Set- Patients with non-estimated number of exacerbations- COPD degree of severity (GOLD group)

| Non-estimated number of exacerbations- COPD degree of severity (GOLD group) | N | % |
|---|---|---|
| А | | |
| В | | |
| С | | |
| D | | |
| Missing | | |
| Patients in FAS with non-estimated number of exacerbations | | |

Final 3.0, 12.03.2019 32 / 53

# Sensitivity analysis- Table 10: Full Analysis Set- Patients with non-estimated number of exacerbations- COPD degree of severity (GOLD group) [grouped]

| Sensitivity analysis II- COPD degree of severity (GOLD group) [grouped] | N | % |
|---|---|---|
| A/B | | |
| C/D | | |
| Missing | | |
| Patients in FAS with non-estimated number of exacerbations | | |

# Sensitivity analysis- Table 11: Full Analysis Set- Patients with non-estimated number of exacerbations- COPD degree of severity (GOLD group) – Distribution

| | | АВ | | С | | D | | Missing | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Sensitivit | Sensitivity analysis II- GOLD stadium- Distribution | % | Ν | % | Z | % | Ν | % | Ν | % |
| Symptoms Exacerbations | | | | | | | | | | |
| 0-1 | 0-1 | | | | | | | | | |
| 0-1 | >=2 | | | | | | | | | |
| 2-4 | 0-1 | | | | | | | | | |
| 2-4 | >=2 | | | | | | | | | |
| Patients in FAS with non-estimated number of exacerbations | | | | | | | | | | |

Sensitivity analysis- Table 12: Full Analysis Set- Patients with non-estimated number of exacerbations- Total CCQ score- Share of patients with therapeutic success after 6 weeks (approximately)- defined as 0.4-point decrease of total CCQ score between baseline and week 6 (approximately)

| *************************************** | CCQ | NI | % | CLOE9/ |
|---|---|---|---|---|
| Sensitivity analysis II- Share | e of patients with therapeutic success | N | % | CI 95% |
| | Therapy successful | | | |
| Gold A | Therapy not successful | | | |
| | Missing | | | |
| | Total | | | |
| | Therapy successful | | | |
| GOLD B | Therapy not successful | | | |
| | Missing | | | |
| | Total | | | |
| | Therapy successful | | | |
| GOLD C | Therapy not successful | | | |
| GOLD C | Missing | | | |
| | Total | | | |
| | Therapy successful | | | |
| GOLD D | Therapy not successful | | | |
| GOLD D | Missing | | | |
| | Total | | | |
| Total | Therapy successful | | | |
| I Ulai | Therapy not successful | | | |

Final 3.0, 12.03.2019 33 / 53

| Sensitivity analysis II- Share | CCQ e of patients with therapeutic success | N | % | CI 95% |
|---|---|---|---|---|
| | Missing | | | |
| | Total | | | |

# Sensitivity analysis- Table 13: Full Analysis Set- Patients with non-estimated number of exacerbations- CCQ score

| | >>> Q000 | ***** | XX | Maga | CL OF9/ | 044 | Min | Modion | Mov | Masiaa |
|---|---|---|---|---|---|---|---|---|---|---|
| Sensiti | ivity analysis II- CC | Q score | N | Mean | CI 95% | Std | Min | Median | Max | Nmiss |
| | | А | | | | | | | | |
| | | В | | | | | | | | |
| | Symptom | С | | | | | | | | |
| | | D | | | | | | | | |
| | | Total | | | | | | | | |
| | | А | | | | | | | | |
| | | В | | | | | | | | |
| | Functional state (CCQ-4) | С | | | | | | | | |
| | State (OOQ-4) | D | | | | | | | | |
| | | Total | | | | | | | | |
| | | Α | | | | | | | | |
| | | В | | | | | | | | |
| | Mental state | С | | | | | | | | |
| | | D | | | | | | | | |
| | | Total | | | | | | | | |
| | | А | | | | | | | | |
| Baseline<br>(Visit 1) | | В | | | | | | | | |
| (VIOIC 1) | Total CCQ score | С | | | | | | | | |
| | 00010 | D | | | | | | | | |
| | | Total | | | | | | | | |
| | | А | | | | | | | | |
| | | В | | | | | | | | |
| | Symptom | С | | | | | | | | |
| | | D | | | | | | | | |
| | | Total | | | | | | | | |
| | | А | | | | | | | | |
| | | В | | | | | | | | |
| | Functional state (CCQ-4) | С | | | | | | | | |
| | 0.0.0 (000 4) | D | | | | | | | | |
| | | Total | | | | | | | | |
| | | А | | | | | | | | |
| | Mental state | В | | | | | | | | |
| | | С | | | | | | | | |

| CCQ | | N | Mean | CI 95% | Std | Min | Median | Max | Nmiss |
|---|---|---|---|---|---|---|---|---|---|
| Sensitivity analysis II- CC | Q score | | | | | | | | |
| | D | | | | | | | | |
| | Total | | | | | | | | |
| | Α | | | | | | | | |
| | В | | | | | | | | |
| Total CCQ score | С | | | | | | | | |
| 30010 | D | | | | | | | | |
| | Total | | | | | | | | |

Final 3.0, 12.03.2019 35 / 53

#### 2.5 Tables for subgroup analysis

#### For each of the following subgroups

- Maintenance naïve patients vs. patients already treated at baseline (i.e. before start of therapy with Spiolto<sup>®</sup> Respimat<sup>®</sup>) with long-acting bronchodilators (LAMA only or LABA only) or LABA+ICS [Only if both categories include more than 20% of all patients, respectively]
- Maintenance naïve patients vs. patients already treated at baseline with long-acting bronchodilators (LAMA only) vs patients already treated at baseline with long-acting bronchodilators (LABA only) vs patients already treated at baseline with long-acting bronchodilators (LABA+ICS)
- ICS treatment at baseline (Patients with ICS vs. Patients without ICS) [Only if both categories include more than 20% of all patients, respectively]
- GOLD spirometric classifications (Group 1) (1/2 vs. 3/4)
- GOLD spirometric classifications (Group 2) (2 vs. 3 vs. 4)
- GOLD patients group (Group 1) (B vs. C/D)
- GOLD patients group (Group 2) (B vs. C vs. D)
- Age (≤ 65 years vs. >65 years)
- Exacerbations in the last 12 months (≤1 vs. ≥2)
- Hospitalizations due to exacerbations (0 vs. ≥1)
- Smoker (Smoker vs. Ex-Smoker vs. Non-smoker)
- Patients with cardiac comorbidities (No vs. Yes)
- Continuation of Spiolto<sup>®</sup> Respimat<sup>®</sup> usage after end of study observation (No vs. Yes)

Table 1 to Table 9 given below will be displayed for each subgroup, respectively, subgroup and group 1, group ... are respective placeholders.

#### Primary endpoints

Subgroup analysis-Table 1: Analysis stratified by subgroup-Full Analysis Set-Total CCQ score-Share of patients with therapeutic success after 6 weeks (approximately), defined as 0.4-point decrease of total CCQ score between baseline and week 6 (approximately)

| co | N | % | CI 95% |
|------------------------|------------------------|----|----------|
| Share of patients with | IN | /0 | CI 93 /6 |
| | Therapy successful | | |
| Group 1 | Therapy not successful | | |
| | Missing | | |
| | Total | | |
| | Therapy successful | | |
| Group | Therapy not successful | | |
| Group | Missing | | |
| | Total | | |
| Total | Therapy successful | | |

Final 3.0, 12.03.2019 36 / 53
| CCQ | | N | % | CI 95% |
|------------------------|------------------------|----|----|----------|
| Share of patients with | therapeutic success | IN | /0 | CI 95 /6 |
| | Therapy not successful | | | |
| | Missing | | | |
| | Total | | | |

# Subgroup analysis- Table 2: Analysis stratified by subgroup- Full Analysis Set- Total CCQ score- Share of patients with therapeutic success- $\chi^2$ -Test (Fisher's Exact test)

| X²-Test (Fisher's Exact test) - Therapy success | p-Value |
|-------------------------------------------------|---------|
| Group 1 vs. Group | |

#### Subgroup analysis- Table 3: Analysis stratified by subgroup- Full Analysis Set- CCQ score

| ************ | >cco>>>>> | XXXXXXX | N | Mean | CI | Std | Min | Median | Max | Nmiss |
|---|---|---|---|---|---|---|---|---|---|---|
| CCQ score | | | | 95% | | | | | | |
| Symptom | | Group 1 | | | | | | | | |
| | Symptom | Group | | | | | | | | |
| | | Total | | | | | | | | |
| | | Group 1 | | | | | | | | |
| | Functional state (CCQ-4) | Group | | | | | | | | |
| Baseline (Visit 1) | otate (CCQ 4) | Total | | | | | | | | |
| | | Group 1 | | | | | | | | |
| | Mental state | Group | | | | | | | | |
| | | Total | | | | | | | | |
| | Total CCQ<br>score | Group 1 | | | | | | | | |
| | | Group | | | | | | | | |
| | 30016 | Total | | | | | | | | |
| | | Group 1 | | | | | | | | |
| | Symptom | Group | | | | | | | | |
| | | Total | | | | | | | | |
| | | Group 1 | | | | | | | | |
| | Functional state (CCQ-4) | Group | | | | | | | | |
| Week 6 (appr.) | State (CCQ-4) | Total | | | | | | | | |
| (Visit 2) | | Group 1 | | | | | | | | |
| | Mental state | Group | | | | | | | | |
| | | Total | | | | | | | | |
| | | Group 1 | | | | | | | | |
| | Total CCQ score | Group | | | | | | | | |
| | 33310 | Total | | | | | | | | |

### Secondary endpoints

# Subgroup analysis- Table 4: Analysis stratified by subgroup- Full Analysis Set- Absolut change of CCQ score between visit 1 and visit 2

| CCQ CCQ score- Change between baseline and Week 6 (approximately) | | N | Mean | CI<br>95% | Std | Min | Median | Max | Nmiss |
|---|---|---|---|---|---|---|---|---|---|
| | Group 1 | | | | | | | | |
| Symptom | Group | | | | | | | | |
| | Total | | | | | | | | |
| | Group 1 | | | | | | | | |
| Functional state (CCQ-4) | Group | | | | | | | | |
| (334 1) | Total | | | | | | | | |
| | Group 1 | | | | | | | | |
| Mental state | Group | | | | | | | | |
| | Total | | | | | | | | |
| | Group 1 | | | | | | | | |
| Total CCQ score | Group | | | | | | | | |
| | Total | | | | | | | | |

# Subgroup analysis- Table 5: Analysis stratified by subgroup- Full Analysis Set- Absolut change of CCQ- Wilcoxon Rank-Sum Test (Mann-Whitney-U-Test)/Kruskal-Wallis Test

| Change from baseline-<br>Wilcoxon Rank-Sum Test (Mann-Whitney-U-Test)/Kruskal-Wallis Test | p-Value |
|---|---|
| CCQ-4 score- Group 1 vs. Group | |
| Total CCQ score- Group 1 vs. Group | |

# Subgroup analysis- Table 6: Analysis stratified by subgroup- Full Analysis Set- General condition of patient (PGE score)

| General condition of patient (PGE score) | | Gro | up 1 | Group | | Total | |
|---|---|---|---|---|---|---|---|
| | | N | % | N | % | N | % |
| anamnesis.general_condition | 1 | | | | | | |
| | 2 | | | | | | |
| | 3 | | | | | | |
| | 4 | | | | | | |
| | 5 | | | | | | |
| Baseline (Visit 1) | 6 | | | | | | |
| | 7 | | | | | | |
| | 8 | | | | | | |
| | Missing | | | | | | |
| | Number of patients | | | | | | |
| visit.general_condition | 1 | | | | | | |
| | 2 | | | | | | |
| Week 6 (approximately) (Visit 2) | 3 | | | | | | |
| | 4 | | | | | | |

Final 3.0, 12.03.2019 38 / 53

| General condition of patient (PGE score) | | Group 1 | | Group | | Total | |
|---|---|---|---|---|---|---|---|
| | | Ν | % | N | % | N | % |
| | 5 | | | | | | |
| | 6 | | | | | | |
| | 7 | | | | | | |
| | 8 | | | | | | |
| | Missing | | | | | | |
| | Number of patients | | | | | | |

<sup>\*</sup>bad=1-2, satisfactory=3-4, good=5-6, excellent=7-8

# Subgroup analysis- Table 7: Analysis stratified by subgroup- Full Analysis Set- General condition of patient (PGE score)- $\chi^2$ -Test

| PGE- X²-Test* | p-Value |
|--------------------------------------------|---------|
| Baseline- Group 1 vs. Group | |
| Week 6 (approximately) - Group 1 vs. Group | |

<sup>\*</sup>If  $\chi^2$ -Test is not valid, Fisher's Exact test will be done or PGE will be treated as continuous variable and compared by Wilcoxon Rank-Sum Test (Mann-Whitney-U-Test)/Kruskal-Wallis Test.

# Subgroup analysis- Table 8: Analysis stratified by subgroup- Full Analysis Set- Patient satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup>

| Patient satisfaction | | Gro | up 1 | Group | | Total | |
|---|---|---|---|---|---|---|---|
| | | N | % | N | % | N | % |
| visit.satisfaction_spiolto | Very satisfied | | | | | | |
| | Satisfied | | | | | | |
| | Rather satisfied | | | | | | |
| | Neither satisfied nor dissatisfied | | | | | | |
| Patient overall | Rather dissatisfied | | | | | | |
| satisfaction with Spiolto® Respimat® treatment | Dissatisfied | | | | | | |
| Respimat <sup>®</sup> treatment | Very dissatisfied | | | | | | |
| | Not answered | | | | | | |
| | Missing | | | | | | |
| | Total | | | | | | |
| visit.satisfaction_inhalator | Very satisfied | | | | | | |
| | Satisfied | | | | | | |
| | Rather satisfied | | | | | | |
| | Neither satisfied nor dissatisfied | | | | | | |
| Patient satisfaction with | Rather dissatisfied | | | | | | |
| inhaling from the | Dissatisfied | | | | | | |
| Respimat <sup>®</sup> device | Very dissatisfied | | | | | | |
| | Not answered | | | | | | |
| | Missing | | | | | | |
| | Total | | | | | | |
| visit.satisfaction_handling | Very satisfied | | | | | | |
| Patient satisfaction with | Satisfied | | | | | | |

Final 3.0, 12.03.2019 39 / 53

| Patient satisfaction | | Group 1 | | Group | | Total | |
|---|---|---|---|---|---|---|---|
| | | N | % | N | % | N | % |
| handling of the Respimat <sup>®</sup> inhalation | Rather satisfied | | | | | | |
| device | Neither satisfied nor dissatisfied | | | | | | |
| | Rather dissatisfied | | | | | | |
| | Dissatisfied | | | | | | |
| | Very dissatisfied | | | | | | |
| | Not answered | | | | | | |
| | Missing | | | | | | |
| | Total | | | | | | |

# Subgroup analysis- Table 9: Analysis stratified by subgroup- Full Analysis Set- Patient satisfaction with Spiolto $^{\!0}$ Respimat $^{\!0}$ - $\chi^2$ -Test

| Satisfaction assessment- X²-Test* | p-Value |
|---|---|
| Patient overall satisfaction with Spiolto® Respimat® therapy- Group 1 vs. Group | |
| Patient satisfaction with inhalation device Respimat®- Group 1 vs. Group | |
| Patient satisfaction with handling of the inhalation device- Group 1 vs. Group | |

<sup>\*</sup>If  $\chi^2$ -Test is not valid, Fisher's Exact test will be done or satisfaction will be treated as continuous variable and compared by Wilcoxon Rank-Sum Test (Mann-Whitney-U-Test)/Kruskal-Wallis Test.

### 2.6 Appendix

## Appendix 1: Other reason for not performing corresponding visit (free text)

| [anamnesis,visit].done_reason_spec | Bas | eline | Visit 2 | |
|---|---|---|---|---|
| Other reason for not performing corresponding visit | N | % | N | % |
| Reason 1 | | | | |
| Reason 2 | | | | |
| Total | | | | |

#### Appendix 2: Other concomitant diseases during observation (free text)

| [anamnesis,visit].disease_other_spec | Baseline | | Visit 2 | |
|--------------------------------------|----------|---|---------|---|
| Other concomitant diseases | N | % | N | % |
| Disease 1 | | | | |
| Disease 2 | | | | |
| Total | | | | |

#### Appendix 3: Concomitant medication during observation (free text)

| [anamnesis,visit]_medication.drug Concomitant medication | N | % |
|-----------------------------------------------------------|---|---|
| Medication 1 | | |
| Medication 2 | | |
| Total | | |

#### Appendix 4: Concomitant medication during observation- Other diseases treated

| [anamnesis,visit]_medication.disease_spc | N % | |
|------------------------------------------------|-----|----|
| Concomitant medication- Other diseases treated | IN | 70 |
| Disease 1 | | |
| Disease 2 | | |
| Total | | |

#### Appendix 5: Other respiratory therapeutics prior/during observation (free text)

| [anamnesis;visit]_resp.therapy_spec | Baseline | Vis | it 2 |
|-------------------------------------|----------|-----|------|
| Other respiratory therapeutics | N % | N | % |
| Therapeutic 1 | | | |
| Therapeutic 2 | | | |
| Total | | | |

Final 3.0, 12.03.2019 41 / 53

#### Appendix 6: Respiratory therapeutics prior/during observation- Trade name (free text)

| [anamnesis,visit]_resp.therapy_spec | Baseline | | Visit 2 | |
|-------------------------------------|----------|---|---------|---|
| Trade name of therapeutic | N | % | N | % |
| Name 1 | | | | |
| Name 2 | | | | |
| Total | | | | |

## Appendix 7: Other reasons for irregular treatment with Spiolto® Respimat® (free text)

| visit.spiolto_regular_reason_spc Other reason for irregular treatment with Spiolto® Respimat® | N | % |
|---|---|---|
| Reason 1 | | |
| Reason 2 | | |
| Total | | |

## Appendix 8: Other reasons for no continuation of Spiolto® Respimat® treatment (free text)

| visit.spiolto_reason_spec Other reason for no continuation of Spiolto® Respimat® treatment | N | % |
|---|---|---|
| Reason 1 | | |
| Reason 2 | | |
| Total | | |

## Appendix 9: Adverse events- No causality with Spiolto®- Suspected context (free text)

| sae.spiolto_causality_spec | N | % |
|-----------------------------------------------|----|----|
| No causality with Spiolto®- Suspected context | 17 | 70 |
| Context 1 | | |
| Context 2 | | |
| Total | | |

## Appendix 10: Adverse events- Other reason for seriousness (free text)

| sae.criteria_other_spec | N | 0/ |
|----------------------------------------------|----|----|
| Adverse events- Other reason for seriousness | IN | % |
| Criteria 1 | | |
| Criteria 2 | | |
| Total | | |

Final 3.0, 12.03.2019 42 / 53

## Appendix 11: Cause of death (free text)

| sae.criteria_other_spec | N | % |
|-------------------------|----|----|
| Cause of death | IN | /0 |
| Cause 1 | | |
| Cause 2 | | |
| Total | | |

Final 3.0, 12.03.2019

43 / 53

### 2.7 Listings

### Listing 1: Patients with visit 1- Violation of inclusion or exclusion criteria (Patients with violations only)

| org. name; org.city | patient.no | | *********** | | *********** |
|---|---|---|---|---|---|
| Site | Patient-No. | Violation of inclusion criteria | Which criteria | Violation of exclusion criteria | Which criteria |

#### Listing 2: Patients with visit 1- Disposition

| org. name; org.city | patient.no | | *********** | | |
|---|---|---|---|---|---|
| Site | Patient-No. | Included in Treated Set | Reason, why not | Included in FAS | Reason, why not |

### **Listing 3: Treated Set- GOLD group**

| org. name;<br>org.city | patient.no | mmrc.act<br>ivity | anamnesis.exacerb ation | anamnesis.estimate | anamnesis.exacerb<br>ation_hospital | anamnesis.estimate_ho<br>spital | <b>****</b> |
|---|---|---|---|---|---|---|---|
| Site | Patient-<br>No. | mMRC<br>classifica<br>tion | Exacerbations<br>within the last 12<br>months before initial<br>visit | Number of exacerbations estimated? | Hospitalizations due to exacerbations | Number of hospitalizations due to exacerbations estimated? | GOLD<br>group |

#### **Listing 4: Treated Set- Patient characteristics**

| org. name;<br>org.city | patient.no | Age | patient.<br>gender | anamnesis.copd_year | anamnesis.spiolto_training |
|---|---|---|---|---|---|
| Site | Patient-No. | Age | Gender | Year of initial COPD diagnosis | Training with Spiolto® Respimat® |

Final 3.0, 12.03.2019 44 / 53

## **Listing 5: Treated Set- Subgroup classification**

| org.<br>name;<br>org.city | patient.<br>no | Age | anamnesis_respiratory;<br>anamnesis_resp.therapy | | anamnesis<br>.copd_<br>severity | | anamn<br>esis.<br>exacer<br>bation | anamnesis.<br>exacerbation_<br>hospital | anam-<br>nesis.<br>smoker | anamnesis.<br>disease_<br>cardiac | anamnesis.<br>spiolto_<br>reason |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Sito | Patient- | <b>A G G</b> | Maintenance ICS | COPD | GOLD | Within the last 12 months before initial visit | | Smoker | Cardiac | Continuation of medication | |
| Site Patient-No. | No. | Ade | naïve/<br>Pretreated | treatment<br>at baseline | degree of severity | group | Exacer-<br>bations | Hospitalizations due to excerbations | Sillokei | comorbidities | after end of observation |

### **Listing 6: Treated Set- Study course (Visit 2)**

| org.<br>name;<br>org.city | patient.<br>no | visit.<br>done | visit.done_<br>reason | visit.spiolto_regular | visit.spiolto_<br>regular_reason | visit.smoker_<br>change | visit.spiolto_<br>pregnancy | visit.spiolto_<br>continued | visit.spiolto_<br>reason |
|---|---|---|---|---|---|---|---|---|---|
| Site | Patient-<br>No. | Visit 2<br>done | Reason why not | Therapy with Spiolto <sup>®</sup><br>Respimat <sup>®</sup> carried out<br>regularly | Reason for irregular treatment | Smoker-<br>Changes in<br>smoking<br>since visit 1 | Pregnancy<br>during<br>treatment | Continuation of medication after end of observation | Reason for discontinuation |

## Listing 7: Treated Set- Concomitant diseases at baseline

| org. name; org.city | patient.no | anamnesis.disease | anamnesis.disease_allergic;; anamnesis.disease_other |
|---|---|---|---|
| Site | Patient-No. | Concomitant diseases | Which disease |

Final 3.0, 12.03.2019 45 / 53

#### Listing 8: Treated Set-Concomitant diseases during study course

| org. name; org.city | patient.no | visit.disease | visit_disease.type ; visit_disease.disease | |
|---|---|---|---|---|
| Site | Patient-No. | Change of concomitant diseases | Existing diagnosis at visit 1 now-defunct | New diagnosis after visit 1 |

#### Listing 9: Treated Set- Concomitant medication at baseline

| org. name; org.city | patient.no | anamnesis.medication | anamnesis_medication.drug | anamnesis_medication.disease |
|---|---|---|---|---|
| Site | Patient-No. | Concomitant medication | Which medication | Disease treated |

## Listing 10: Treated Set- Concomitant medication during study course

| org. name; org.city | patient.no | visit.disease | visit_me | edication.type; visit_medica | tion.disease; visit_medicat | ion.drug |
|---|---|---|---|---|---|---|
| Site | Patient-No. | Change of concomitant medciation | Existing medication at visit 1 discontinued since then- Medication | Existing medication at visit 1 discontinued since then- Disease treated | New medication after visit 1- Medication | New medication after visit 1- Disease treated |

#### Listing 11: Treated Set- Treatment with past COPD therapies (Patients with past COPD therapies only)

| org. name; org.city | patient.no | anamnesis.respiratory | anamnesis_resp.therapy | anamnesis_resp.name | anamnesis_resp.prescribe |
|---|---|---|---|---|---|
| Site | Patient-No. | Treatment with past COPD therapies | Therapeutics | Trade name | Prescription |

## Listing 12: Treated Set- Treatment with other COPD related therapies besides Spiolto® Respimat® during study course

| org. name; org.city | patient.no | visit.disease | visit_resp.type ; vis | it_resp.therapeutic |
|---|---|---|---|---|
| Site | Patient-No. | Change of other COPD related therapies besides Spiolto® | Components of existing baseline therapy at visit 1 discontinued since then | New therapy in addition to already existing baseline therapies besides Spiolto® Respimat® introduced after visit 1 |

Final 3.0, 12.03.2019 46 / 53

### Listing 13: Full Analysis Set- CCQ – Primary endpoint

| org. name; org.city | patient.no | | ccq.q_01-ccq.q_10 | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Detient No | | | В | asel | ine- | Que | stion | ıs | | | Visit 2- Questions | | | | | | | |
| | Patient-No. | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 |

### Listing 14: Full Analysis Set- Primary and secondary endpoint- Therapeutic success and change between baseline and Visit 2

| org.<br>name;<br>org.city | patient. | | | | | | | ccq.q_01- | ccq.q_10 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Patient- | Symptom | symptom (Q1; Q2; Q5; Q6) Functional state (CCQ-4) (Q7-Q10) Mental state (Q3; Q4) Tot | | | | | | Total CC | otal CCQ score | | | | | |
| Sile | No. | Baseline | Visit 2 | Change | Baseline | Visit 2 | Change | Success | Baseline | Visit 2 | Change | Baseline | Visit 2 | Change | Success |

#### Listing 15: Full Analysis Set- Secondary endpoints

| org. name;<br>org.city | patient.<br>no | anamnesis.<br>general_condition | visit.general_<br>condition | visit.satisfaction_spiolto | visit.satisfaction_inhalator | visit.satisfaction_handling |
|---|---|---|---|---|---|---|
| Site | Patient-<br>No. | Baseline- PGE score | Week 6 (appr.)-<br>PGE score | Patient overall satisfaction with Spiolto <sup>®</sup> Respimat <sup>®</sup> treatment | Patient satisfaction with inhaling from the Respimat® device | Patient satisfaction with handling of the Respimat <sup>®</sup> inhalation device |

### Listing 16: Treated Set - Drug-related adverse events

| org.<br>name;<br>org.city | patient.no | Age | patient.<br>gender | sae.nci | Coded by | Coded by | sae.start; anamnesis.<br>spiolto_date; visit.date;<br>visit.spiolto_last_date | sae.<br>start | sae.<br>end | sae.therapy | sae.<br>outcome | sae.spiolto_<br>action_taken | sae.sae |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Patient-<br>No. | Age | Sex | Event | SOC term | PT term | Point in time* | Start<br>date | End<br>date | Therapy required | Outcome | Action taken | Serious? |

Final 3.0, 12.03.2019 47 / 53

Listing 17: Treated Set - Serious adverse events

| org.<br>name;<br>org.city | patient.<br>no | Age | patient.<br>gender | sae.nci | Coded<br>by | Coded<br>by | sae.start; anamnesis.<br>spiolto_date; visit.date;<br>visit.spiolto_last_date | sae.<br>start | sae.<br>end | sae.<br>outcome | sae.spiolto<br>_causality | sae.spiolto_<br>action_taken | sae.criteria_[fatal; life_<br>threatening; disability;<br>hospital; prolonged;<br>congenital; other] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Patient-<br>No. | Age | Sex | Event | SOC<br>term | PT<br>term | Point in time* | Start<br>date | End<br>date | Outcome | Relation | Action taken | Reason |

<sup>\*</sup> Point in time  $\in$  {Screening; Treatment; Post-treatment}

## Listing 18: Treated Set - Cause of death

| org. name; org.city | patient.no | Age | patient.gender | sae.death_date | sae.death_cause |
|---|---|---|---|---|---|
| Site | Patient-No. | Age | Sex | Date of death | Cause of death |

Final 3.0, 12.03.2019 48 / 53

#### **Tables**

```
Table 15.1.1 1: Disposition
```

Table 15.1.2 1: Patients with visit 1- Important protocol violations

Table 15.1.2 2 Patients with visit 1- Inclusion criteria

Table 15.1.2 3: Patients with visit 1- Exclusion criteria

#### Table 15.1.3 1: Patients with visit 1 patients- Summary of analysis population

Table 15.1.4 1: Treated Set- Age at registration [years]

Table 15.1.4 2: Treated Set- Age at registration, categorical

Table 15.1.4 3: Treated Set- Gender

Table 15.1.4 4: Treated Set- Height [cm]

Table 15.1.4 5: Treated Set- Weight [kg]

Table 15.1.4 6: Treated Set- Duration between initial diagnosis of COPD and baseline visit [years]

Table 15.1.4 7: Treated Set- COPD degree of severity (spirometric)

Table 15.1.4 8: Treated Set- COPD degree of severity (spirometric) [grouped]

#### Table 15.1.4 9: mMRC Questionnaire

Table 15.1.4 10: Treated Set- Exacerbations and hospitalizations due to excerbations in the last 12 months

Table 15.1.4 11: Treated Set- Exacerbations and hospitalizations due to excerbations in the last 12 months, categorical

Table 15.1.4 12: Treated Set- COPD degree of severity (GOLD group)

Table 15.1.4 13: Treated Set- COPD degree of severity (GOLD group) [grouped]

Table 15.1.4 14: Treated Set- COPD degree of severity (GOLD group) – Distribution

Table 15.1.4 15: Treated Set- COPD degree of severity (GOLD group) - Smoking

Table 15.1.4 16: Treated Set- COPD degree of severity (GOLD group) – ICS at baseline

Table 15.1.4 17: Treated Set- Patients with concomitant diseases

Table 15.1.4 18: Treated Set- Concomitant diseases (multiple answers possible)

Table 15.1.4 19: Treated Set- Concomitant diseases- Gastrointestinal/Hepatobiliary (multiple answers possible)

Table 15.1.4 20: Treated Set- Concomitant diseases- Pulmonary (except COPD) (multiple answers possible)

Table 15.1.4 21: Treated Set- Concomitant diseases- Metabolic/Endocrine (multiple answers possible)

Table 15.1.4 22: Treated Set- Concomitant diseases- Muscular-skeletal/ Dermatological (multiple answers possible)

Table 15.1.4 23: Treated Set- Smoking

Table 15.1.4 24: Treated Set- Smoking- Pack-years

Table 15.1.4 25: Treated Set- Patients with concomitant medication (except respiratory therapeutics)

Table 15.1.4 26: Treated Set- Diseases treated with concomitant medication (except respiratory therapeutics)- (multiple answers possible)

Table 15.1.4 27: Treated Set- Concomitant medication (except respiratory therapeutics)- Continuation or new prescription (multiple answers possible)

Table 15.1.4 28: Treated Set-Spiolto® Respirat® - Patient trained to use inhaler

Table 15.1.4 29: Treated Set- Treatment with past COPD therapies (6 weeks prior to start of study treatment) according to mMRC value

- Table 15.1.4 30: Treated Set- Treatment with past COPD therapies (6 weeks prior to start of study treatment)- Respiratory therapeutics (multiple answers possible)
- Table 15.1.4 31: Treated Set- Therapy with Spiolto<sup>®</sup> Respimat<sup>®</sup> carried out regularly
- Table 15.1.4 32: Treated Set- Reason for therapy with Spiolto<sup>®</sup> Respimat<sup>®</sup> carried out irregularly
- Table 15.1.4 33: Treated Set- Changes of treatment with other COPD related therapies besides Spiolto<sup>®</sup> Respimat<sup>®</sup> since visit 1 [i.e. new therapy introduced or existing baseline therapy discontinued\*]
- Table 15.1.4 34: Treated Set- Changes of treatment with other COPD related therapies besides Spiolto<sup>®</sup> Respimat<sup>®</sup> since visit 1- Affected respiratory therapeutics (multiple answers possible)
- Table 15.1.4 35: Treated Set- Changes of concomitant diseases since visit 1 [i.e. new diagnosis or now-defunct diagnosis]
- Table 15.1.4 36: Treated Set- Changes of concomitant diseases- Diseases (multiple answers possible)
- Table 15.1.4 37: Treated Set- Changes of concomitant medication since visit 1 [i.e. new medication introduced or existing medication discontinued]
- Table 15.1.4 38: Treated Set- Changes of concomitant medication- Disease treated
- Table 15.1.4 39: Treated Set- Smokers at baseline- Current status (smoking status at visit 2)
- Table 15.1.4 40: Treated Set- Pregnancy during treatment
- Table 15.2.1 1: Full Analysis Set- Total CCQ score- Share of patients with therapeutic success after 6 weeks (approximately), defined as 0.4-point decrease of total CCQ score between baseline and week 6 (approximately)
- Table 15.2.1 2: Full Analysis Set- CCQ score
- Table 15.2.1 3: Full Analysis Set- Absolut change of CCQ score between baseline and week 6 (approximately)
- Table 15.2.1 4: Full Analysis Set- General condition of the patient evaluated by the physician (PGE- score)
- Table 15.2.1 5: Full Analysis Set- Patient satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup>
- Table 15.3.1 1: Treated Set- Time between start of treatment and end of observation/discontinuation [weeks]
- Table 15.3.1 2: Treated Set- Survival status
- Table 15.3.2 1: Treated Set- Adverse events overall summary
- Table 15.3.2 2: Treated Set- Drug-related AE according to MedDRA-SOC and PT (event based)
- Table 15.3.2 3: Treated Set- Drug-related AE by MedDRA system organ class and preferred term- Maximum NCI grade per patient
- Table 15.3.2 4: Treated Set- Number of patients with drug-related AE occurring with share in preferred term greater than 5% by primary system organ class and preferred term
- Table 15.3.2 5: Treated Set- Drug-related AE- Worst outcome per patient
- Table 15.3.2 6: Treated Set- Drug-related AE- Patients with at least one drug-related AE for which therapy was required

50 / 53

- Table 15.3.2 7: Treated Set- Drug-related AE- Patient pregnant at AE
- Table 15.3.2 8: Treated Set- Drug-related AE- Week of pregnancy
- Table 15.3.2 9: Treated Set- Drug-related AE- Action taken concerning therapy (patient based; multiple answers possible)

Final 3.0, 12.03.2019

- Table 15.3.2 10: Treated Set- Drug-related AE leading to treatment discontinuation by MedDRA system organ class and preferred term
- Table 15.3.2 11: Treated Set- Drug-related AE- Improvement after stop of therapy (patient based; multiple answers possible)
- Table 15.3.2 12: Treated Set- Drug-related AE- Re-exposition done for at least one event
- Table 15.3.2 13: Treated Set- Drug-related AE- Recurrence of at least one TEAE after re-exposition
- Table 15.3.2 14: Treated Set- Incorrect administration of medication (multiple answers possible)
- Table 15.3.2 15: Treated Set- Serious AE according to MedDRA-SOC and PT (event based)
- Table 15.3.2 16: Treated Set- Serious AE- Reason for seriousness (patient based; multiple answers possible)
- Table 15.3.2 17: Treated Set- Serious AE by MedDRA system organ class and preferred term- Maximum NCI grade per patient
- Table 15.3.2 18: Treated Set- Serious AE- Worst outcome per patient
- Table 15.3.2 19: Treated Set- Serious AE- Action taken concerning treatment (patient based; multiple answers possible)
- Table 15.3.2 20: Treated Set- Serious AE leading to treatment discontinuation by MedDRA system organ class and preferred term
- Table 15.3.2 21: Treated Set- Serious AE- Number of patients with at least one serious AE with causal relationship to treatment
- Table 15.3.2 22: Treated Set- Serious AE by relationship with Spiolto<sup>®</sup> Respimat<sup>®</sup> by MedDRA system organ class and preferred term

#### Sensitivity analyses

- Sensitivity analysis- Table 1: Full Analysis Set- Time between Visit 1 and Visit 2 [weeks]
- Sensitivity analysis- Table 2: Full Analysis Set- Time between Visit 1 and Visit 2 [categorical]
- Sensitivity analysis- Table 3: Analysis stratified by time between Visit 1 and Visit 2- Full Analysis Set- Total CCQ score- Share of patients with therapeutic success after 6 weeks (approximately)- defined as 0.4-point decrease of total CCQ score between baseline and week 6 (approximately)
- Sensitivity analysis- Table 4: Analysis stratified by time between Visit 1 and Visit 2-Full Analysis Set- Total CCQ score- Share of patients with therapeutic success- $\chi^2$ -Test (Fisher's Exact test)
- Sensitivity analysis- Table 5: Analysis stratified by time between Visit 1 and Visit 2-Full Analysis Set- CCQ score
- Sensitivity analysis- Table 6: Full Analysis Set- Patients with non-estimated number of exacerbations
- Sensitivity analysis- Table 7: Full Analysis Set- Patients with non-estimated number of exacerbations- Exacerbations in the last 12 months
- Sensitivity analysis- Table 8: Full Analysis Set- Patients with non-estimated number of exacerbations- Exacerbations in the last 12 months [categorical]
- Sensitivity analysis- Table 9: Full Analysis Set- Patients with non-estimated number of exacerbations- COPD degree of severity (GOLD group)
- Sensitivity analysis- Table 10: Full Analysis Set- Patients with non-estimated number of exacerbations- COPD degree of severity (GOLD group) [grouped]

51 / 53

Final 3.0, 12.03.2019

- Sensitivity analysis- Table 11: Full Analysis Set- Patients with non-estimated number of exacerbations- COPD degree of severity (GOLD group) Distribution
- Sensitivity analysis- Table 12: Full Analysis Set- Patients with non-estimated number of exacerbations- Total CCQ score- Share of patients with therapeutic success after 6 weeks (approximately)- defined as 0.4-point decrease of total CCQ score between baseline and week 6 (approximately)
- Sensitivity analysis- Table 13: Full Analysis Set- Patients with non-estimated number of exacerbations- CCQ score

#### Subgroup analyses

- Subgroup analysis- Table 1: Analysis stratified by subgroup- Full Analysis Set- Total CCQ score- Share of patients with therapeutic success after 6 weeks (approximately), defined as 0.4-point decrease of total CCQ score between baseline and week 6 (approximately)
- Subgroup analysis- Table 2: Analysis stratified by subgroup- Full Analysis Set- Total CCQ score- Share of patients with therapeutic success-  $\chi^2$ -Test (Fisher's Exact test)
- Subgroup analysis- Table 3: Analysis stratified by subgroup- Full Analysis Set- CCQ score
- Subgroup analysis- Table 4: Analysis stratified by subgroup- Full Analysis Set-Absolut change of CCQ score between visit 1 and visit 2
- Subgroup analysis- Table 5: Analysis stratified by subgroup- Full Analysis Set-Absolut change of CCQ- Wilcoxon Rank-Sum Test (Mann-Whitney-U-Test)/Kruskal-Wallis Test
- Subgroup analysis- Table 6: Analysis stratified by subgroup- Full Analysis Set-General condition of patient (PGE score)
- Subgroup analysis- Table 7: Analysis stratified by subgroup- Full Analysis Set-General condition of patient (PGE score)-  $\chi^2$ -Test
- Subgroup analysis- Table 8: Analysis stratified by subgroup- Full Analysis Set-Patient satisfaction with Spiolto<sup>®</sup> Respirat<sup>®</sup>
- Subgroup analysis- Table 9: Analysis stratified by subgroup- Full Analysis Set-Patient satisfaction with Spiolto<sup>®</sup> Respimat<sup>®</sup>-  $\chi^2$ -Test

#### **Appendix**

- Appendix 1: Other reason for not performing corresponding visit (free text)
- Appendix 2: Other concomitant diseases during observation (free text)
- Appendix 3: Concomitant medication during observation (free text)
- Appendix 4: Concomitant medication during observation- Other diseases treated
- Appendix 5: Other respiratory therapeutics prior/during observation (free text)
- Appendix 6: Respiratory therapeutics prior/during observation- Trade name (free text)
- Appendix 7: Other reasons for irregular treatment with Spiolto<sup>®</sup> Respimat<sup>®</sup> (free text)
- Appendix 8: Other reasons for no continuation of Spiolto® Respimat® treatment (free text)
- Appendix 9: Adverse events- No causality with Spiolto®- Suspected context (free text)
- Appendix 10: Adverse events- Other reason for seriousness (free text)
- Appendix 11: Cause of death (free text)

#### Listings

Listing 1: Patients with visit 1- Violation of inclusion or exclusion criteria (Patients with violations only)

- Listing 2: Patients with visit 1- Disposition
- Listing 3: Treated Set- GOLD group
- Listing 4: Treated Set- Patient characteristics
- Listing 5: Treated Set- Subgroup classification
- Listing 6: Treated Set- Study course (Visit 2)
- Listing 7: Treated Set- Concomitant diseases at baseline
- Listing 8: Treated Set- Concomitant diseases during study course
- Listing 9: Treated Set- Concomitant medication at baseline
- Listing 10: Treated Set- Concomitant medication during study course
- Listing 11: Treated Set- Treatment with past COPD therapies (Patients with past COPD therapies only)
- Listing 12: Treated Set-Treatment with other COPD related therapies besides Spiolto<sup>®</sup> Respimat<sup>®</sup> during study course
- Listing 13: Full Analysis Set- CCQ Primary endpoint
- Listing 14: Full Analysis Set- Primary and secondary endpoint- Therapeutic success and change between baseline and Visit 2
- Listing 15: Full Analysis Set- Secondary endpoints
- Listing 16: Treated Set Drug-related adverse events
- Listing 17: Treated Set Serious adverse events
- Listing 18: Treated Set Cause of death